CLINICAL TRIAL: NCT05907408
Title: Precision Medicine in Fatty Liver Disease: How to Identify the Patient Who Develops Steatohepatitis Using Omics Techniques
Brief Title: Omics Techniques in Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Guilherme Rezende, Associate Professor, Universidade Federal do Rio de Janeiro
Other Study IDs: NASHOmics1
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: nonalcoholic fat liver disease; NASH; metabolic fat liver disease; risk factors; noninvasive markers; transcriptomics; metabolomics; proteomics; liver fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steatosis: Patients with non-alcoholic fatty liver disease presenting exclusively with steatosis, without fibrosis or inflammation
- Steatohepatitis: Patients with non-alcoholic fatty liver disease presenting with steatosis and degree >1 of liver fibrosis

SUMMARY:
Nonalcoholic steatohepatitis (NASH) is the most common cause of chronic liver disease in Western countries and one of the leading causes of liver transplantation in the world. Its spectrum ranges from simple steatosis to decompensated cirrhosis, resulting from progressive fibrosis due to inflammation and cellular injury. The reasons why patients with the same degree of steatosis have different evolutions are not sufficiently known. The objective of this project is to identify biomarkers that predict disease progression, using omics techniques, which can serve to develop new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome
* Liver steatosis detected on transient hepatic elastography performed in the last 12 months
* Steatosis with or without fibrosis confirmed histologically in a liver biopsy performed in the last 12 months

Exclusion Criteria:

* Concurrent liver disease (other than NAFLD)
* Chronic or prolonged use of any potential hepatotoxic drug or substance
* HIV infection
* Cancer (except basal cell carcinoma)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Quaternary university hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Steatosis, without fibrosis or inflammation | 12 months
  Patients with non-alcoholic fatty liver disease presenting exclusively with steatosis, without fibrosis or inflammation
Steatohepatitis, with fibrosis | 12 months
  Patients with non-alcoholic fatty liver disease presenting with steatosis and degree >1 of liver fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme FM Rezende, MD PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.